CLINICAL TRIAL: NCT03460444
Title: Impact of Raising B-OHB Directly With MCT Oil on NLPR3 Inflammasome Activation in Healthy, Young Adults
Brief Title: The Effect of Raising Ketones Directly With MCT Oil on Inflammation in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H17-03258
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: MCT Oil Supplementation
Keywords: NLR Family, Pyrin Domain-Containing 3 Protein; Caspase 1; 3-Hydroxybutyric Acid; Histone Deacetylase Inhibitors; MCT Oil

STUDY DESIGN:
Intervention Model Description: All participants complete the supplementation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCT Oil Supplementation (Experimental): Participants consume MCT oil (97-99% octanoic acid) twice per day for 14 days while consuming a diet similar to the recommended health guidelines (40-50% carbohydrate; 30-40% fat; 20-25% protein).
  Interventions: Dietary Supplement: MCT Oil Supplementation

INTERVENTIONS:
Dietary Supplement: MCT Oil Supplementation — Participants consume MCT oil (97-99% octanoic acid) twice per day for 14 days. Dosing will begin at 5ml/dose for Days 1-2, 10ml for Days 3-4, and 15ml for the remainder of the intervention.

SUMMARY:
Ketogenic diets are gaining support as a method to lower inflammation within the body, but studies have not been able to show the way by which this occurs. Ketones, which are molecules made by the body as a source of energy during carbohydrate restriction, have been shown to have the ability to alter the number and types of messages that immune cells send to each other, and thus have the potential to lower inflammation. To determine whether raising ketones independent of diet reduce inflammation, 20 healthy, young men and women will follow a 14-day "normal" diet combined with MCT oil supplements. Based on previous research, the investigators expect that raising ketones will reduce immune cell pro-inflammatory signaling.

DETAILED DESCRIPTION:
The potential for a ketogenic diet to reduce inflammation has become increasingly popular in recent years, but direct scientific evidence to demonstrate that ketones impact inflammatory mechanisms in humans does not exist. B-hydroxybutyrate (B-OHB) is the most abundant circulating ketone and recent evidence indicates that B-OHB may be able to act as a direct signal to inhibit cellular pathways involved in inflammation.

B-OHB can be raised naturally by induction of nutritional ketosis, which is a normal physiological response to severe reductions in carbohydrate or caloric intake. In this state, free fatty acids are converted to ketone bodies (primarily B-hydroxybutyrate [B-OHB]) by the liver in order to provide essential fuel for metabolically active tissues. However, determining the direct effects of B-OHB in human ketogenic diet studies is difficult due to the numerous metabolic adaptations that occur in nutritional ketosis (e.g., reduced insulin, elevated free fatty acids, stable glucose) and the propensity for participants to lose body and fat mass over longer period.

B-OHB can also be raised independent of diet by supplementation with medium chain triglyceride (MCT) oil, allowing for induction of ketosis without the additional metabolic adaptations. In addition to being an important fuel source, recent interest has focused on a potential signaling role for B-OHB with cell culture and animal studies describing anti-inflammatory, anti-oxidant, and anti-cancer effects. The cellular pathways through which B-OHB is proposed to reduce inflammation, include the NLPR3 inflammasome and histone deacetylases (HDACs), both of which play important roles in regulating cellular inflammation. The NLRP3 inflammasome pathway is an immune complex which, upon activation, initiates downstream pro-inflammatory cascades including the activation of caspase-1 and interleukin (IL)-1B. These pro-inflammatory cascades have been implicated in the propagation of sterile inflammation, which has been identified as a major contributor to certain chronic inflammatory diseases such as type 2 diabetes and atherosclerosis. HDACs are enzymes typically found within the nucleus and have the ability to regulate signaling through innate immune pathways. B-OHB has been shown to have the ability to inhibit HDACs, and consequently has the potential to decrease oxidative stress and inflammation. The NLRP3 inflammasome and HDACs are responsive to the intracellular nutritional milieu and thus their activity may be able to be modulated through increases in B-OHB.

The use of MCT oil supplements will allow the investigators to raise blood B-OHB independent of diet, and thus directly test the immunomodulatory effects of B-OHB in healthy, adult males. This fundamental research is needed to understand whether ketones have direct immunomodulatory effects or if it is the widespread systemic metabolic adaptation to a ketogenic diet that might impact inflammatory processes.

The overall objective of this pilot study is to determine if directly raising B-OHB through supplementation with MCT oil impacts innate immune cell function and/or phenotype. Based on previous cell culture and animal research showing that B-OHB can reduce pro-inflammatory signaling, it is hypothesized that raising B-OHB with MCT oil supplementation will result in a attenuation of caspase-1 activation and mature IL-1B secretion, both markers of NLRP3 inflammasome activation. Additionally, it is hypothesized that raised B-OHB will result in greater histone acetylation, as B-OHB has been shown to be an HDAC inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-29.9 kg/m^2
* Females only: have a regular 28-35 day menstrual cycle

Exclusion Criteria:

* Diagnosed metabolic disorder such as diabetes, metabolic syndrome, hypothyroidism, or any other condition known to affect metabolism;
* history of inflammatory disorders such as Rheumatoid Arthritis, Crohn's Disease, Irritable Bowel Syndrome
* Prescribed any anti-inflammatory medication cannot be avoided for the duration of the study;
* current consumption of a very low-carbohydrate diet (e.g., "Atkins", "Protein Power Plan", "Paleo diet", etc.) or have within the previous three months;
* adhere to dietary restrictions such as vegetarianism or veganism;
* unable to abstain from drugs (prescription and recreational) or alcohol for the duration of the study;
* competitive athlete (currently training for an elite sport).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Caspase-1 Activation at 14 days | Measured the day before the first dose of MCT oil (baseline) and the last day of the 14 day trial (post).
  Caspase-1 activation will be quantified by flow cytometry. The fluorescent inhibitor probe FAM-YVAD-FMK binds covalently to activated caspase-1 and emits at 530nm.

SECONDARY OUTCOMES:
Change from Baseline Histone H3 Acetylation at 14 days | Measured the day before the first dose of MCT oil (baseline) and the last day of the 14 day trial (post).
  Histone H3 acetylation status will be quantified by flow cytometry using the conjugated acetyl-histone H3 antibody specific for Lys9 (Pacific Blue 455) and the conjugated acetyl-histone H3 antibody specific for Lys14 (Alexa Fluor 488).
Change from Baseline Interleukin(IL)-1beta at 14 days | Measured the day before the first dose of MCT oil (baseline) and the last day of the 14 day trial (post).
  Mature IL-1beta secretion will be quantified by enzyme-linked immunosorbent assay run in duplicate.
Change from Baseline Blood beta-hydroxybutyrate at 14 days | Measured the day before the first dose of MCT oil (baseline), 1 and 2 hours after each meal on Day 1, 2, 13, and 14, as well as once every 2 days at a time which is convenient for the participant (i.e. on Day 4, 6, 8, 10, & 12).
  Blood beta-hydroxybutyrate will be quantified in whole blood using FreeStyle Precision Blood β-Ketone Test Strips (Abbott, Abbot Park, IL, USA) with the FreeStyle Precision Neo Blood Ketone Monitoring System (Abbott).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No